CLINICAL TRIAL: NCT04439903
Title: Web-Based Simulation Tool For Self-Management Support In Type 1 Diabetes Mellitus
Acronym: WST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Research Associate, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200157
Record Dates: First submitted 2020-06-14; First posted 2020-06-19 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
Keywords: Web-based Simulation Tool (WST); Continuous Glucose Monitoring (CGM); Glucose Metabolism Model; Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single-arm, single center, non-randomized, uncontrolled pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based Simulation Tool (WST) (Experimental)
  Interventions: Other: Web-based Simulation Tool

INTERVENTIONS:
Other: Web-based Simulation Tool — Glucose, insulin and meal data from the participants' insulin pump will be collected and entered into the WST, which will generate personalized models of the participants' glucose metabolism to enable replay simulations.

SUMMARY:
This project focuses on embedding the participants' own diabetes data into state-of-the-art technology platforms to constitute a novel educational simulation interface for decision-support in Type 1 Diabetes (T1D) - the Web-based Simulation Tool (WST).

DETAILED DESCRIPTION:
The Web-based Simulation Tool (WST) allows patients with Type 1 Diabetes (T1D) to not only visualize their data, but also to explore changes to their meals and insulin parameters, and easily estimate their potential clinical impact. WST is an educational tool, and as such, it does not have prescriptive power. This platform collects glucose, insulin and meal data from the participants' insulin pump, and generates personalized models of their glucose metabolism. Both data collection and model personalization are backend processes, that is, without user intervention.

Participants can interact with WST through a user interface (UI) that is equipped with a dashboard page, where they can:

(i) select a particular date range using a calendar to visualize their historical glucose control, such as glucose traces, and time in range;

(ii) control the amount of information on the screen - users can show/hide more details, such as glucose variability;

(iii) select different insulin therapy parameters: basal rate, insulin sensitivity factor, and carbohydrate ratio;

(iv) change their values by moving a slider;

(v) select informed meals within the selected date range, and modify their time and size by moving a slider;

(vi) run a simulation with the modified insulin therapy parameters and meals by tapping a button;

(vii) save the insulin and meal settings of the simulations to compare multiple configurations; and

(viii) generate a report from the selected simulation, comparing both original and simulated or replay data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 and ≤65 years old at time of consent.
* Clinical diagnosis, based on investigator assessment, of T1D for at least one year.
* Using insulin for at least 1 year prior to study enrollment.
* Using an insulin pump for at least 6 months prior to study enrollment.
* Currently using a CGM for at least 6 months.
* Willingness to use a Dexcom G6 CGM during the study; a study Dexcom CGM will be provided if needed.
* Current user of the Tandem t:slim X2 insulin pump.
* Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study.
* Total daily insulin (TDI) dose at least 10 U/day.
* HbA1c ≤9.0% at screening; if HbA1c <6.0%, then TDI must be ≥ 0.5 U/kg.
* Having access to internet (Wi-Fi or 3G, 4G, 5G, or similar).
* Willingness to interact with a computer program.
* An understanding of and willingness to follow the protocol and sign the informed consent form (ICF).

Exclusion Criteria:

* Participants who are not able to read and complete questionnaires on the computer or interact with a program for which they will be trained because of language, reading, or cognitive issues.
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment.
* History of a seizure disorder (except hypoglycemic seizure), unless written clearance is received from a neurologist and not currently on a seizure medication.
* Pregnancy, breast-feeding, or intention of becoming pregnant over time of study procedures.
* If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.
* A known medical condition that in the judgment of the investigator might interfere with the completion of the study.*
* Abuse of alcohol or recreational drugs.
* Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis, etc).
* Uncontrolled arterial hypertension (resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg).
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol.
* Current use of the following drugs and supplements:

  * Any drug other than insulin to treat diabetes.
  * Any other medication that according to the investigator's criteria is a contraindication for the subject's participation.

    * Note: The software implementation, in the current development status, is designed to interact with subjects with T1D that only use insulin for diabetes treatment and do not present any comorbidity related to diabetes.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Colmegna, PhD, Principal Investigator — University of Virginia, Center for Diabetes Technology
Locations (1):
- University of Virginia - Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- [Background] Colmegna P, Bisio A, McFadden R, Wakeman C, Oliveri MC, Nass R, Breton M. Evaluation of a Web-Based Simulation Tool for Self-Management Support in Type 1 Diabetes: A Pilot Study. IEEE J Biomed Health Inform. 2023 Jan;27(1):515-525. doi: 10.1109/JBHI.2022.3209090. Epub 2023 Jan 4. PMID 36149995
- [Result] Colmegna P, McFadden R, Fabris C, Lobo B, Nass R, Oliveri MC, Brown SA, Kovatchev B. Adaptive Biobehavioral Control: A Pilot Analysis of Human-Machine Coadaptation in Type 1 Diabetes. Diabetes Technol Ther. 2024 Sep;26(9):644-651. doi: 10.1089/dia.2023.0399. Epub 2024 Apr 30. PMID 38662425

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Web-based Simulation Tool (WST)
Started | 18
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 1
  Unknown or Not Reported | 0
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — Population: 1 participant did not meet inclusion criteria, and 2 participants withdrew for scheduling purposes prior to Hemoglobin A1c measurement.
  Percentage of glycosylated hemoglobin
    number analyzed (Participants) | 15
    (all) | 6.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Technology Expectation and Technology Acceptance Questionnaires: Perceived Burdens and Benefits at Baseline and Week 5 (Post-intervention)
Description: Technology Expectation (TE) and Technology Acceptance (TA) questionnaires are made of 27 items. Responses to the TE questionnaire were collected at week 0 (baseline), and responses to the TA questionnaire at week 5 (post-intervention). Each questionnaire has 5 categories: burdens (14 items), benefits (10 items), ease of use, usefulness, and trustworthiness (last 3, 1 item each). Items are scored on a 5-point Likert scale ranging from 1 to 5 (from strongly disagree to strongly agree for burdens and benefits, and from very poor to excellent for ease of use, usefulness, and trustworthiness). Here we report the results for burdens and benefits. The original 1-to-5 scale is converted to a 0-to-4 scale, the mean scores for burdens and benefits are averaged and then converted into a percentage ranging from 0% to 100%. Higher percentages mean a better outcome for benefits and a worse outcome for burdens.
Time Frame: Baseline and Week 5 (Post-intervention)
Measure: Median (Inter-Quartile Range); unit: percentage of mean item score
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 15
percentage of mean item score
  Burdens_Baseline | 25.0 [14.4 to 38.1]
  Burdens_Post-intervention | 42.5 [21.3 to 51.3]
  Benefits_Baseline | 58.9 [52.7 to 68.8]
  Benefits_Post-intervention | 55.4 [38.4 to 66.1]

2. Primary Outcome: Technology Expectation and Technology Acceptance Questionnaires: Perceived Ease of Use, Usefulness and Trustworthiness of the System at Baseline and Week 5 (Post-intervention)
Description: Technology Expectation (TE) and Technology Acceptance (TA) questionnaires are made of 27 items. Responses to the TE questionnaire were collected at week 0 (baseline), and responses to the TA questionnaire at week 5 (post-intervention). Each questionnaire has 5 categories: burdens (14 items), benefits (10 items), ease of use, usefulness, and trustworthiness (last 3, 1 item each). Items are scored on a 5-point Likert scale ranging from 1 to 5 (from strongly disagree to strongly agree for burdens and benefits, and from very poor to excellent for ease of use, usefulness, and trustworthiness). Here we report the results for ease of use, usefulness, and trustworthiness of the system. Higher scores mean a better outcome.
Time Frame: Baseline and Week 5 (Post-intervention)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 15
score on a scale
  ease-of-use_Baseline | 4 [3 to 4]
  ease-of-use_Post-intervention | 3 [3 to 4]
  usefulness_Baseline | 4 [4 to 4]
  usefulness_Post-intervention | 4 [3 to 4]
  trustworthiness_Baseline | 4 [4 to 4]
  trustworthiness_Post-intervention | 4 [3 to 4]

3. Secondary Outcome: Diabetes Distress Scale at Baseline and Week 5 (Post-intervention)
Description: The Diabetes Distress Scale (DDS) is a 17-item scale that yields a total diabetes distress score plus 4 subscale scores: Emotional burden (5 items), regimen distress (5 items), interpersonal distress (3 items) and physician distress (4 items). Scores range from 1 to 6 (from Not a problem to A very serious problem). To compute the total diabetes distress score and the 4 subscale scores, participants' responses in each scale are summed and divided by the corresponding number of items. A mean item score lower than 2.0 is considered little or no distress, between 2.0 and 2.9 is considered moderate distress, and higher than 3.0 is considered high distress. Thus, higher scores mean a worse outcome.
Time Frame: Baseline and Week 5 (Post-intervention)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 15
score on a scale
  Total-Diabetes-Distress_Baseline | 1.9 [1.5 to 2.0]
  Total-Diabetes-Distress_Post-intervention | 1.8 [1.3 to 2.4]
  Emotional-Burden_Baseline | 2.2 [1.7 to 3.4]
  Emotional-Burden_Post-intervention | 2 [1.7 to 2.4]
  Regimen-Distress_Baseline | 1.6 [1.4 to 2.5]
  Regimen-Distress_Post-intervention | 1.4 [1.2 to 2.3]
  Interpersonal-Distress_Baseline | 2 [1.2 to 2.6]
  Interpersonal-Distress_Post-intervention | 2 [1.1 to 2.6]
  Physician-Distress_Baseline | 1 [1 to 1.2]
  Physician-Distress_Post-intervention | 1 [1 to 1]

4. Other Pre Specified Outcome: Potential Correlation Between System Use and Changes in the Percentage of Time Spent in 70-180 mg/dL Between First Week (Observation) and Following 4 Weeks (Intervention)
Description: The percentage of time spent in 70-180 mg/dL (time in range, TIR) is computed per participant on a weekly basis (1 week of observation, 4 weeks of intervention) using glucose sensor data. The higher the TIR the better the glucose control. Percentages during the intervention period are averaged per participant, thus obtaining 2 TIRs for each participant (one Observation TIR and one Intervention TIR). A linear regression analysis is performed to infer the impact (if any) of the duration and frequency of participants' interaction with the Web-Based Simulation Tool (predictor variables) on variations in TIR between Observation and Intervention periods (response variable).
  Predictor variable 1: Number of simulations per participant per week. Predictor variable 2: Minutes of interaction with the Web-Based Simulation Tool per participant per week.
  Response variable: Intervention TIR - Observation TIR. The higher the response variable the better the outcome.
Time Frame: First Week (Observation) and Following 4 Weeks (Intervention)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 15
percentage of time | -0.8 (5.8)
Statistical Analysis 1: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.61532, Regression, Linear; Intercept = 1.9726, Standard Error of Mean 3.8238
Statistical Analysis 2: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.5128, Regression, Linear; Slope = -0.68016, Standard Error of Mean 1.0084 — Predictor variable 1: Number of simulations per participant per week
Statistical Analysis 3: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.68197, Regression, Linear; Slope = 0.15238, Standard Error of Mean 0.3629 — Predictor variable 2: Minutes of interaction with the Web-Based Simulation Tool per participant per week

5. Other Pre Specified Outcome: Potential Correlation Between System Use and Changes in Perceived Regimen Distress at Baseline and Week 5 (Post-intervention)
Description: Perceived regimen distress is estimated at Baseline and Week 5 (Post-intervention) using the Diabetes Distress Scale (DDS). Scores range from 1 to 6 (from Not a problem to A very serious problem). Participants' responses to the DSS's regimen distress items are summed and divided by the number of items in that scale. Higher scores mean a worse outcome. Scores at week 5 are compared with scores at baseline and used in a linear regression analysis to infer the impact (if any) of the duration and frequency of participants' interaction with the Web-Based Simulation Tool (predictor variables) on variations in treatment satisfaction (response variable).
  Predictor variable 1: Number of simulations per participant per week. Predictor variable 2: Minutes of interaction with the Web-Based Simulation Tool per participant per week.
  Response variable: Regimen distress score at week 5 - Regimen distress score at baseline. The higher the response variable the worse.
Time Frame: Baseline and Week 5 (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 15
score on a scale | -0.17 (0.71)
Statistical Analysis 1: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.28789, Regression, Linear; Intercept = -0.49527, Standard Error of Mean 0.44535
Statistical Analysis 2: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.17848, Regression, Linear; Slope = 0.16785, Standard Error of Mean 0.11745 — Predictor variable 1: Number of simulations per participant per week
Statistical Analysis 3: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.17514, Regression, Linear; Slope = -0.06091, Standard Error of Mean 0.042266 — Predictor variable 2: Minutes of interaction with the Web-Based Simulation Tool per participant per week

6. Other Pre Specified Outcome: Potential Correlation Between System Use and Changes in Perceived Emotional Burden at Baseline and Week 5 (Post-intervention)
Description: Perceived emotional burden is estimated at Baseline and Week 5 (Post-intervention) using the Diabetes Distress Scale (DDS). Scores range from 1 to 6 (from Not a problem to a very serious problem). Participants' responses to the DSS's emotional burden items are summed and divided by the number of items in that scale. Higher scores mean a worse outcome. Scores at week 5 are compared with scores at baseline and used in a linear regression analysis to infer the impact (if any) of the duration and frequency of participants' interaction with the Web-Based Simulation Tool (predictor variables) on variations in treatment satisfaction (response variable).
  Predictor variable 1: Number of simulations per participant per week. Predictor variable 2: Minutes of interaction with the Web-Based Simulation Tool per participant per week.
  Response variable: Emotional burden score at week 5 - Emotional burden score at baseline.
  The higher the response variable the worse.
Time Frame: Baseline and Week 5 (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Simulation Tool (WST)
Number analyzed (Participants) | 15
score on a scale | -0.33 (0.934)
Statistical Analysis 1: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.63929, Regression, Linear; Intercept = -0.28825, Standard Error of Mean 0.59949
Statistical Analysis 2: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.37964, Regression, Linear; Slope = -0.14422, Standard Error of Mean 0.1581 — Predictor variable 1: Number of simulations per participant per week
Statistical Analysis 3: Comparison: Web-based Simulation Tool (WST); Test type: Other; p = 0.26057, Regression, Linear; Slope = 0.06718, Standard Error of Mean 0.056895 — Predictor variable 2: Minutes of interaction with the Web-Based Simulation Tool per participant per week

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Web-based Simulation Tool (WST)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Web-based Simulation Tool (WST) (N=15)
COVID positive (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The Tandem t:connect web application was down for one month due to maintenance work, affecting considerably 4 participants who did not have the opportunity to interact with up-to-date data during a significant part of Phase 2 (system-use phase).

No data was excluded in computing the outcomes, despite this issue (and the COVID positive case).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT04439903/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT04439903/ICF_001.pdf